CLINICAL TRIAL: NCT07160075
Title: Improving Access to HIV Pre-exposure Prophylaxis: Implementation and Evaluation of Innovative HIV Prevention Services Among Persons on Opioid Replacement Therapy in Western Canada: Prospective, Implementation Study
Brief Title: HIV Prevention With PrEP Among People on Opioid Replacement Therapy
Acronym: OAT-PrEP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cara Spence (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Cara Spence, Lead Principal Investigator in Saskatchewan, Canada, University of Saskatchewan
Organization: University of Saskatchewan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Bio 5418
Record Dates: First submitted 2025-08-18; First posted 2025-09-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: HIV - Human Immunodeficiency Virus
Keywords: PrEP; OAT; Opioid Agonist Therapy; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Group (Experimental): Participants who have agreed to be on PrEP
  Interventions: Behavioral: Simultaneous administration of OAT and oral PrEP at existing pharmacy-based programs
- Non-PrEP Group (No Intervention): Participants who have declined PrEP

INTERVENTIONS:
Behavioral: Simultaneous administration of OAT and oral PrEP at existing pharmacy-based programs — Simultaneous administration of OAT and oral PrEP (direct observed therapy or home supply) at existing pharmacy-based programs
  Arms: PrEP Group

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of providing oral pre-exposure prophylaxis (PrEP) and opioid agonist therapy (OAT) simultaneously in existing pharmacy-based programs operating in Alberta and Saskatchewan, to collect preference, adherence, and persistence data on oral PrEP, and to assess interest / acceptability of long-lasting injectable options for human immunodeficiency virus (HIV) prevention.

DETAILED DESCRIPTION:
In Alberta and Saskatchewan, Canada, HIV acquisition is increasingly and predominantly seen in people who inject drugs (PWID). Less than 2% of this population are utilizing PrEP despite a high level of new infections. The purpose of this study is to assess the feasibility and acceptability of providing oral PrEP and OAT simultaneously in existing pharmacy-based programs operating in Alberta and Saskatchewan, to collect preference, adherence, and persistence data on oral PrEP, and to assess interest and acceptability of long-lasting injectable options for HIV prevention.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative
* Ongoing behaviors with potential HIV exposure as assessed by a clinician
* Regularly engaged with their respective OAT program at least 3 days a week for the past 2 weeks
* Report willingness to return for follow-up visits

Exclusion Criteria:

* Creatine clearance <30 mL/min or any medical condition or medication known to be contraindicated with the use of Emtricitabine/Tenofovir Alafenamide (F/TAF) or Emtricitabine/Tenofovir Disoproxil Fumarate (F/TDF)
* Taken PrEP within the last 24 hours at the time of screening or enrollment
* Deemed appropriate by a clinician for HIV Post-Exposure Prophylaxis at the time of screening or enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Oral PrEP use in an OAT setting at 6 months follow-up: Review data from participant screening and clinical follow-up, and compare it to baseline PrEP use to assess uptake | Start of 6-month recruitment period to 6 months following the end of the recruitment period
  The proportion of participants:
  * Using PrEP within the clinical programs at baseline
  * Who initiate PrEP (take one dose) when approached for study enrollment and 1, 3, and 6 months from study initiation
  * Maintained on PrEP at 6 months (have taken PrEP at least once a week)
Oral PrEP use in an OAT setting at 6 months follow-up: Record the time from offer to acceptance of PrEP | From the time that PrEP was offered to the acceptance of PrEP or the end of the 6-month recruitment period

SECONDARY OUTCOMES:
Compare usage and clinical outcomes between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  PrEP adherence data will be collected via self-report and dispensing records (daily direct observed therapy and pill count for home supply).
  Unit of measure for PrEP adherence: Number of weeks in which PrEP prescription was filled.
  The proportion of participants adhering to PrEP will be compared between the PrEP and non-PrEP arms.
Compare usage and clinical outcomes between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  OAT adherence through self-report and dispensing records (daily direct observed therapy and pill count for home supply)
Compare usage and clinical outcomes between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Overall persistence, i.e.: PrEP taken at least once per week
Compare usage and clinical outcomes between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Overall persistence, i.e.: OAT taken at least once per week
HIV incidence between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
STI incidence between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
Compare usage and clinical outcomes between individuals who initiate PrEP and those who do not at 1, 3, 6, 9, and 12 months | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Comparing the number of individuals lost to follow-up between both groups
To determine the barriers, facilitators, preferences, and contextual factors for uptake, adherence, and continuance of PrEP by participants, as well as patient-reported outcome (PRO) measures | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Qualitative measures assessed in all patient participants at baseline, 1, 3, 6, 9, and 12 months: HIV PrEP Stigma Scale (HPSS-12)
  Higher total scores reflect a higher level of perceived HIV-related stigma. Total scores range from 12 to 48.
To determine the barriers, facilitators, preferences, and contextual factors for uptake, adherence, and continuance of PrEP by participants, as well as PRO measures | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Qualitative measures assessed in all patient participants at baseline, 1, 3, 6, 9, and 12 months: Depression Scale (PHQ-9)
  Total scores range from 0 to 27. 0-4 indicates minimal or no depression, 5-9 suggests mild depression, 10-14 indicates moderate depression, 15-19 represents moderately severe depression, and 20-27 signifies severe depression.
To determine the barriers, facilitators, preferences, and contextual factors for uptake, adherence, and continuance of PrEP by participants, as well as PRO measures | From initiation of PrEP to 1, 3, 6, 9, and 12 months after initiation
  Qualitative measures assessed in all patient participants at baseline, 1, 3, 6, 9, and 12 months: Generalized Anxiety Disorder (GAD-7)
  Total scores are interpreted on a scale from 0 to 21, with higher scores indicating more severe anxiety.
To determine the barriers, facilitators, preferences, and contextual factors for uptake, adherence, and continuance of PrEP by participants, as well as PRO measures | At initiation of PrEP
  Qualitative measures will be assessed at baseline by interviewing OAT provider participants with questions regarding awareness of PrEP, barriers and facilitators of PrEP use, preferences for and acceptability of long-acting injectable options.
  Interview questions at Baseline visit:
  * Before this study, how often would you recommend PrEP to patients at risk of HIV?
  * What do you think most of your patients' understanding of PrEP is?
  * Based on your estimates, what proportion of patients with HIV exposure are on PrEP in this community?
  * Why do you think is/are the reason(s) an eligible patient would decline PrEP?
  * In your experience, what are some effective ways to encourage eligible patients to take PrEP?
  * Do you believe health system barriers limit the uptake of PrEP in patients at risk of HIV? If so, what are they?
  * What are your opinions on prescribing a long-acting injectable option for PrEP over the oral version?
To determine the barriers, facilitators, preferences, and contextual factors for uptake, adherence, and continuance of PrEP by participants, as well as PRO measures | 1, 3, 6, 9, and 12 months after initiation of PrEP
  Qualitative measures will be assessed at 1, 3, 6, 9, and 12 months, by interviewing OAT provider participants with questions regarding awareness of PrEP, barriers and facilitators of PrEP use, preferences for and acceptability of long-acting injectable options.
  Interview questions at Follow-up visit:
  * Do you think your patients' understanding of PrEP has changed since the study began? If so, how?
  * Do you think your patients' attitudes towards PrEP has changed since the study began? If so, how?
  * What proportion of your patients do you predict will continue taking PrEP after the study ends? Why?
  * Have your opinions changed on prescribing long-acting injectables for PrEP over the oral version? If so, what is your current opinion and why?
  * Since the last questionnaire, do you have any additional comments on the patient-level and health system-level barriers and facilitators for PrEP uptake in this community?

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Sheldon M Chumir Health Centre, Calgary, Alberta
  - Queen City Wellness Pharmacy, Regina, Saskatchewan
  - Mayfair Drugs Pharmacy, Saskatoon, Saskatchewan
  - Pharmasave Riversdale Pharmacy, Saskatoon, Saskatchewan
  - The Medicine Shoppe Pharmacy, Saskatoon, Saskatchewan
  - Meadowgreen Pharmacy, Saskatoon, Saskatchewan